CLINICAL TRIAL: NCT03695471
Title: A Phase II, Open-Label, Single-Arm Trial Using KEYTRUDA (Pembrolizumab) as Initial Systemic Therapy in the Treatment of Advanced Mycosis Fungoides
Brief Title: Pembrolizumab in Treating Patients With Stage IB-IV Mycosis Fungoides
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1788; NCI-2018-02023 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17-010349 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2018-10-02; First posted 2018-10-04 (Actual); Results first posted 2025-08-11 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2024-12

CONDITIONS: Mycosis Fungoides; Sezary Syndrome; Stage IB Mycosis Fungoides and Sezary Syndrome AJCC v8; Stage II Mycosis Fungoides and Sezary Syndrome AJCC v8; Stage IIA Mycosis Fungoides and Sezary Syndrome AJCC v8; Stage IIB Mycosis Fungoides and Sezary Syndrome AJCC v8; Stage III Mycosis Fungoides and Sezary Syndrome AJCC v8; Stage IIIA Mycosis Fungoides and Sezary Syndrome AJCC v8; Stage IIIB Mycosis Fungoides and Sezary Syndrome AJCC v8; Stage IV Mycosis Fungoides and Sezary Syndrome AJCC v8; Stage IVA1 Mycosis Fungoides and Sezary Syndrome AJCC v8; Stage IVA2 Mycosis Fungoides and Sezary Syndrome AJCC v8; Stage IVB Mycosis Fungoides and Sezary Syndrome AJCC v8
MeSH Terms: conditions — Mycosis Fungoides; Sezary Syndrome | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (pembrolizumab) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 24 cycles or until complete response in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II trial studies how well pembrolizumab works in treating patients with stage IB-IV mycosis fungoides. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the antitumor activity of pembrolizumab in patients with advanced mycosis fungoides (MF) as initial systemic therapy.

SECONDARY OBJECTIVES:

I. To evaluate safety of pembrolizumab in this patient population. II. To evaluate response rates of pembrolizumab in this patient population. III. To determine the progression free survival, duration of response, time to response and overall survival of pembrolizumab in this patient population.

CORRELATIVE OBJECTIVE:

I. To characterize the histologic features of the anti-tumor response in patients with advanced MF before and after treatment with pembrolizumab.

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Treatment repeats every 21 days for up to 24 cycles or until complete response in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 and 90 days, and then every 3 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Histological confirmation of one of the following:

  * Stage IIB-IV mycosis fungoides not previously treated with systemic therapy
  * Stage IB/IIA mycosis fungoides with Modified Severity Weighted Assessment Tool (mSWAT) >= 20 with high risk morphologic features defined as thick plaque disease and/or follicular involvement who have failed one form of skin-directed therapy.
  * Sezary syndrome patients not previously treated with systemic therapy.
* Measurable disease based on mSWAT and/or Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Note: Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to registration. Exception: Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the Sponsor.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1.
* Absolute neutrophil count (ANC) >= 1,500 /mcL (obtained =< 28 days prior to registration)
* Platelet count >= 100,000/mcL (obtained =< 28 days prior to registration)
* Hemoglobin >= 9.0 g/dL or >= 5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment)
* Serum total bilirubin =< 1.5 X upper limit of normal (ULN) OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN (obtained =< 28 days prior to registration)
* Aspartate transaminase (AST) and alanine transaminase (ALT) =< 2.5 X ULN OR =< 5 X ULN for subjects with liver metastases (obtained =< 28 days prior to registration)
* Albumin > 2.5 mg/dL (obtained =< 28 days prior to registration)
* Serum creatinine =< 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance >= 60 ml/min for subject with creatinine levels > 1.5 x institutional ULN (obtained =< 28 days prior to registration)
* Prothrombin time (PT)/international normalized ratio (INR) and partial thromboplastin time (PTT) =< 1.5 X ULN OR if patient is receiving anticoagulant therapy and PT/INR or PTT is within therapeutic range of intended use of coagulants (obtained =< 28 days prior to registration)
* Negative urine or serum pregnancy test done =< 28 days prior to registration and =< 72 hours prior to receiving the first dose of study medication, for women of childbearing potential only.
* Female subjects of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of the study medication.

  * Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
* Male subjects of childbearing potential must agree to use an adequate method of contraception for the course of the study through 120 days after the last dose of the study medication.

  * Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
* Provide written informed consent.
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study).
* Willing to provide tissue samples for correlative research purposes.

Exclusion Criteria:

* Any of the following because this study involves: an agent that has known genotoxic, mutagenic and teratogenic effects:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Is currently participating and receiving study therapy or have participated in a study of an investigational agent and received study therapy or used an investigational device =< 4 weeks prior to registration.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy =< 7 days prior to registration.
* Has a known history of active TB (Bacillus tuberculosis).
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) =< 4 weeks prior to registration or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy =< 2 weeks prior to registration or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent.

  * Note: Subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study.
  * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions: basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Exceptions: subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging =< 4 weeks prior to registration and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least =< 7 days prior to registration. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Note: Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a history of non-infectious pneumonitis that required steroids or has current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies).
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or Hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected).
* Has received a live vaccine =< 30 days prior to registration.

  * Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed.
* Sezary syndrome patients with high blood burden requiring immediate cytoreduction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2024-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason C. Sluzevich, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Pembrolizumab)
Started | 9
Completed | 8
Not Completed | 1
Not completed — Cancellation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (12.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Overall Cutaneous Responders at Their 9th or Final Cycle (Cutaneous Complete Response [CR], Cutaneous 90 Response [CR90] or Cutaneous Partial Response [PR])
Description: Will be assessed by the Modified Severity Weighted Assessment Tool (mSWAT). All calculated values will use the last-observation-carried forward for any participants who withdraw, are lost to follow up, or exit the study per protocol. The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients will be analyzed using Mann-Whitney U for nonparametric data and the student t-test. Confidence intervals for the true success proportion will be calculated according to the approach of Duffy and Santner. mSWAT is calculated using body surface area (BSA) of each MF lesion (palm plus fingers of the patient ≈ 1% BSA) in each of 12 areas of the body, multiplying the sum of the BSA of each lesion type by a weighting factor (patch=1, plaque=2, and tumor =4) and generating a sum of the subtotals of each lesion subtype.
Time Frame: 7 months
Measure: Number; unit: proportion of participants
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 8
proportion of participants | 0.25

2. Secondary Outcome: Incidence of Adverse Events
Description: The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. The count of participants for each maximum reported adverse event is below.
Time Frame: 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 9
Participants
  Grade 1 | 5
  Grade 2 | 4

3. Secondary Outcome: Percentage Change in mSWAT Score
Description: The Modified Severity-Weighted Assessment Tool (mSWAT) is used to evaluate the extent and severity of skin involvement in mycosis fungoides. It is used to standardize the assessment of skin lesions. A higher mSWAT score indicates greater extent of skin involvement. The total body surface area (BSA) affected by each type of lesion (patches, plaques, and tumors) is estimated, and each lesion type is assigned a weighting factor: patches *1, plaques *2, and tumors *4. The BSA for each lesion type is multiplied by its corresponding weighting factor, and then the weighted values are summed to produce the final mSWAT score. mSWAT is calculated using body surface area (BSA) of each MF lesion (palm plus fingers of the patient ≈ 1% BSA) in each of 12 areas of the body, multiplying the sum of the BSA of each lesion type by a weighting factor (patch=1, plaque=2, and tumor =4) and generating a sum of the subtotals of each lesion subtype.
Time Frame: Baseline to 7 months
Measure: Median (Full Range); unit: Percent change from baseline
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 8
Percent change from baseline | -5.015 [-97.86 to 675.19]

4. Secondary Outcome: Progression Free Survival
Description: The distribution of progression-free survival will be estimated using the method of Kaplan-Meier. In addition, the progression-free survival rate at 5 years after registration will be reported.
Time Frame: 28 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 8
Months | 8.9 [3.4 to NA] — Too few events, upper limit is not calculable.

5. Secondary Outcome: Duration of Response
Description: The distribution of duration of complete response will be estimated using the method of Kaplan-Meier.
Time Frame: 26 months
Population: All evaluable patients that achieved a response during treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 3
Months | 7.6 [2.7 to NA] — Too few events, upper limit is not calculable.

6. Secondary Outcome: Time to Response
Description: Median time to response is defined as the time from registration to CR, CR90 or PR.
Time Frame: 7 months
Population: All evaluable patients that achieved CR, CR90 or PR are included in the analysis. This includes one patient that was not a success for the primary endpoint due to progressing prior to their 9th cycle of treatment.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 3
months | 2.04 [1.38 to 2.23]

7. Secondary Outcome: Median Overall Survival Time
Description: The distribution of survival time will be estimated using the method of Kaplan-Meier. It's defined as the time from a patients registration until death or lost to followup.
Time Frame: 728 days
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 8
months | 10.6 [4.8 to NA] — Not enough events occurred; upper limit is not calculable.

8. Other Pre Specified Outcome: Biomarker Analysis - CD4 Pre and Post Pembrolizumab
Description: Immunohistochemistry will be used to quantify levels of CD4 before and after treatment with pembrolizumab
Time Frame: Up to 1 year
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Biomarker Analysis - CD4 Baseline to Cycle 2
Description: Immunohistochemisty will be used for change in baseline calculations of CD4 at baseline and end of cycle 2
Time Frame: Up to 1 year
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Biomarker Analysis - CD8 Baseline to Cycle 2
Description: Immunohistochemisty will be used for change in baseline calculations of CD8 at baseline and end of cycle 2
Time Frame: Up to 1 year
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Biomarker Analysis - PD-1/CD279 Baseline to Cycle 2
Description: Immunohistochemisty will be used for change in baseline calculations of PD-1/CD279 at baseline and end of cycle 2
Time Frame: Up to 1 year
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Biomarker Analysis - PD-1 Baseline to Cycle 2
Description: Immunohistochemisty will be used for change in baseline calculations of PD-1 at baseline and end of cycle 2
Time Frame: Up to 1 year
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Biomarker Analysis - PD-1 Qualitative
Description: Qualitative measures of the strength of PD-1 expression will use published standardized grading scales for categorical classification purposes.
Time Frame: Up to 1 year
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Biomarker Analysis - CD8 Pre and Post Pembrolizumab
Description: Immunohistochemistry will be used to quantify levels of CD8 before and after treatment with pembrolizumab.
Time Frame: Up to 1 year
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Biomarker Analysis - PD-1/CD279 Pre and Post Pembrolizumab
Description: Immunohistochemistry will be used to quantify levels of PD-1/CD279 before and after treatment with pembrolizumab
Time Frame: Up to 1 year
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Biomarker Analysis - PD-L1 Pre and Post Pembrolizumab
Description: Immunohistochemistry will be used to quantify levels of PD- L1 expression before and after treatment with pembrolizumab
Time Frame: Up to 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 7 months and mortality 30 months so far
Arm/Group | Treatment (Pembrolizumab)
All-Cause Mortality (participants affected / at risk) | 1/8
Serious Adverse Events (participants affected / at risk) | 1/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pembrolizumab) (N=8)
Fungemia (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Erythroderma (Skin and subcutaneous tissue disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pembrolizumab) (N=8)
Constipation (Gastrointestinal disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 3 (6)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 5 (18)
Skin infection (Infections and infestations) | 1 (1)
Creatinine increased (Investigations) | 5 (12)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 1 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (10)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (34)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 2 (3)
Hypertension (Vascular disorders) | 7 (31)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-30): https://cdn.clinicaltrials.gov/large-docs/71/NCT03695471/Prot_SAP_000.pdf
  • Informed Consent Form (2023-08-18): https://cdn.clinicaltrials.gov/large-docs/71/NCT03695471/ICF_001.pdf